## A MOBILE HEALTH INTERVENTION TO INCREASE UPTAKE OF PRENATAL CARE IN SYRIAN REFUGEE POPULATION IN TURKEY

Informed Consent Form

Protocol Idenfitication Number: HeraInc 07/28/2021

## INFORMED CONSENT FORM

## The name of the research:

A Mobile Health intervention to increase uptake of prenatal care in Syrian refugee population in Turkey

**Research supervisor:** Dr. Aral Sürmeli, Medical Search and Rescue Association. +90 535 314 0179, <a href="mailto:a.surmeli@medak.org.tr">a.surmeli@medak.org.tr</a>

Dear participant,

You have been invited to participate in the aforementioned research, which has been planned within the Medical Search and Rescue Association. Before accepting to participate in this research, you must understand the purpose of the research and make your decision freely within the framework of this information. Please read the information below carefully, ask our teammates if you have questions please ask at any point.

The research you will participate in has 2 purposes. The first is to collect information and data on the use of prenatal health services of the Syrian refugee population living in Istanbul, and the second is to understand the effect of mobile phone reminders on the use of prenatal care services.

If you agree to participate in the study, you will be asked to fill in a form about your demographic and health information, participate in a 15-minute training, and download the HERA application to your phone. After signing the consent form, a colleague from the research team will ask you questions about yourself, current pregnancy, previous pregnancies, and other health issues.

After answering the questions, you will attend a briefing session that will take approximately 15 minutes about the HERA application, which is considered as an intervention tool in the research. Please share with our teammates if you have any questions during the session or while filling the form. After the briefing session, you will be asked to download the HERA application to your smartphone. HERA, with reference to your last menstrual day, it will calculate the dates of your least four prenatal medical appointments and age of your pregnancy. You will be reminded of these appointment dates later via the HERA application via notification. Your 4 minimum antenatal care appointments will be reminded to you 3 times: 2 weeks before the appointment date calculated by the HERA system, 1 day before and on the day of the appointment. After the appointment date has passed, you will be asked about whether you have attended the appointment via the HERA application, and if you have not, you will be asked to explain the reason for not

going. This process will continue throughout your pregnancy. At the end of the 6 months, one of our teammates will contact you by phone and ask questions about your appointments.

A total of 162 participants will be included in the research, and you will be expected to spend about 1 hour in total during the 6-month period.

The current research does not pose any risk. Once you have agreed to participate in the research, you have the right not to continue the research. Your participation in the research will not provide you any financial gain or cause any financial loss.

The information collected through the form will be stored in a closed cabinet in the researcher's office, and the information collected through HERA will be stored on a secure server and not shared with anyone outside of the researchers. Only the research supervisor has access to these data. The data collected from you will be made available to the rest of the research team after your personal information (e.g. your name) has been extracted and anonymized.

Taking part in this research is entirely at your discretion. You can refuse to take part in the research or quit after it begins. The results of this research will be used for scientific purposes. If you withdraw from the study or are excluded from the research by the researcher, your data will not be used. **However, once the data is anonymized, you will not be able to withdraw from the research.** All information obtained from you will be kept confidential, and the confidentiality of your identity information, if any, will be protected when the research is published.

I have read (or listened to) the above text, which contains the information that should be given to the volunteers before starting the research. I asked the researchers my questions on issues I thought were missing and got clear answers. I am of the opinion that I understood all the written and oral statements submitted to me in detail. Ample time was given to decide whether I would like to participate in the study.

Under these circumstances, I declare that I accept with my own free will, without any pressure or coercion, the use of my personal information obtained within the scope of the research for scientific purposes, its presentation and publication in compliance with the confidentiality rules. A copy of the consent form is also given to me.

If you prefer not to take part in this study, would you please tell us why below?